CLINICAL TRIAL: NCT04248335
Title: Physiologic Determinants of PPI Disposition in Children
Brief Title: Effect of Obesity on Proton Pump Inhibitors
Acronym: LiverLabPPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kate Kyler, MD, MSc, Physician Scientist, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000201; K23DK115827-01A1 (NIH)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Obesity; NAFLD; GERD
MeSH Terms: conditions — Pediatric Obesity; Non-alcoholic Fatty Liver Disease; Gastroesophageal Reflux | interventions — Pantoprazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- In Weight Management Program (Experimental): Evaluate the effect of liver fat on pharmacology of PPI's, and if applicable midazolam
  Interventions: Drug: Pantoprazole; Drug: Midazolam injection
- Not in Weight Management Program (Experimental): Evaluate the effect of liver fat on drug metabolism of PPI's, and if applicable midazolam
  Interventions: Drug: Pantoprazole; Drug: Midazolam injection

INTERVENTIONS:
Drug: Pantoprazole — single-dose administration
Drug: Midazolam injection — single-dose administration

SUMMARY:
This longitudinal study tests the hypothesis that obesity affects drug pharmacology of acid suppression medications in children.

DETAILED DESCRIPTION:
The purpose of this research study is to see how the body breaks down certain medicines. Many medicines are broken down in the liver. The liver is an organ in the belly. A person's age, size, genetics (DNA), and the health of their liver decide how quickly the body breaks down medicines and how much medication a person needs to take. Everybody's liver has some fat in it, but the amount of fat is different from person to person. The purpose of this study is to see if the amount of fat in the liver affects how quickly acid suppression medications start and stop working and get removed from the body.

ELIGIBILITY:
Inclusion Criteria:

* 6-21 years of age
* Obese and non-obese individuals

  * BMI ≥10th percentile for age (6-20 years of age)
  * BMI ≥18.5 (>20 years of age)
* Otherwise healthy; or otherwise healthy with diagnosis of GERD, NAFLD, chronic abdominal pain or obesity, according to report of medical history and/or review of the medical record
* Receiving or not receiving pantoprazole or lansoprazole for routine medical care
* MRI Hoop Test Clearance

Exclusion Criteria:

* Unable or unwilling to give written permission/assent/consent
* For PO Study Drug: Any anatomic abnormality of the GI tract as defined by history, PE, or radiographic findings, including Bariatric surgery, Nissen fundoplication or equivalent surgery.
* For IV Study Drug: Any anatomic abnormality of the GI tract as defined by history, PE, or radiographic findings, except Bariatric surgery, Nissen fundoplication or equivalent surgery.
* For subjects undergoing weight management, treatment in the last 7 days with proton pump inhibitors omeprazole, esomeprazole, dexlansoprazole, or grapefruit juice.
* For subjects not undergoing weight management, treatment in the last 7 days with medications known to clinically significantly inhibit (e.g., omeprazole, esomeprazole, fluoxetine, fluvoxamine, ketoconazole, ticlopidine, felbamate, trazodone, valproic acid, topiramate) or induce (e.g., phenobarbital, carbamazepine, phenytoin) CYP2C19; and those known at therapeutic doses to significantly inhibit (e.g., erythromycin, clarithromycin, grapefruit juice, verapamil, diltiazem, cimetidine, ketoconazole) or induce (e.g., oxcarbazepine, carbamazepine, phenytoin, phenobarbital, St. John's Wort, rifampin, rifapentine) or CYP3A4 activity in the last 7 days.
* Unable to have blood drawn for the screening lab tests
* Unable or unwilling to fast overnight prior to the study session
* Unable to have blood drawn for the screening lab tests
* If taking lansoprazole or pantoprazole for clinical purposes, unable or unwilling to abstain from that PPI for 3 days prior to PK visit when the PPI is not the same as the study drug for that PK visit
* Metal in the body or any foreign bodies that precludes MRI sequencing
* Claustrophobia
* Exceeds 500lbs or 227 kg in Body Weight
* Demonstrated adverse reaction to previous pantoprazole or PPI exposure
* Impaired hepatic activity as determined by routine liver function testing and defined as values ≥ 5 times the age-specific upper limit of normal (ULN) for AST, ALT, total bilirubin >2.0mg/dl, alkaline phosphatase ≥ 5 times the age-specific ULN
* Impaired renal function defined as creatinine ≥ 3 times the age-specific ULN
* Females of child-bearing age who are pregnant or breast-feeding
* Any known infection with hepatitis B, C, or human immunodeficiency virus (HIV)

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
plasma pharmacokinetics of pantoprazole | 5 years
  plasma maximum peak concentration (Cmax)
plasma pharmacokinetics of pantoprazole | 5 years
  area under the concentration time curve (AUC)
plasma pharmacokinetics of pantoprazole | 5 years
  time to maximum peak concentration (tmax)
plasma pharmacokinetics of pantoprazole | 5 years
  half-life (t 1/2)
plasma pharmacokinetics of pantoprazole | 5 years
  volume of distribution (Vd)
plasma pharmacokinetics of pantoprazole | 5 years
  clearance (CL)

SECONDARY OUTCOMES:
pharmacodynamics | 5 years
  concentration of gastric acid using pH probe test
safety of pantoprazole: incidence of reported and gastrointestinal adverse events | 5 years
  incidence of reported and gastrointestinal adverse events
pharmacokinetics of midazolam, if medication received to ease discomfort of pH probe study | 5 years
  plasma concentrations of midazolam
urinary metabolites | 5 years
  urine concentrations of pantoprazole and midazolam and their metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kyler, MD, MS, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified experimental data may be shared with institutional collaborators outside of CMH and if it is determined that biological samples obtained from study participants must be transferred to institutions outside of CMH for the purpose of confirmatory analyses, appropriate inter-institutional material transfer agreements will first be executed. As this is a pediatric study, minimal blood volumes are being collected and we do not anticipate that biological samples will be available to share with the outside community upon completion of the study, beyond those samples that may be required for confirmatory analyses.